CLINICAL TRIAL: NCT06792357
Title: Effects of Vagus Nerve Stimulation Based on Polyvagal Theory on Labor Pain, Anxiety, Oxytocin, Cortisol Levels, Labor Duration and Perception
Brief Title: Vagus Nerve Stimulation and Labor
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cukurova University (Other)
Responsible Party: Principal Investigator, Rukiye Sülü Dursun, Rukiye Sülü Dursun, Cukurova University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CukurovaUnv; Project NO: 124S403 (Other Grant/Funding Number: TÜBİTAK 1002 - FAST SUPPORT PROGRAM)
Record Dates: First submitted 2024-12-21; First posted 2025-01-24 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: 36-40 haftalık Hamile
Keywords: Emek; oksitozin; kortizol; vagus sinir stimülasyonu; Ebe

STUDY DESIGN:
Intervention Model Description: This project aimed to determine the effect of vagus nerve stimulation based on Polyvagal theory on labor pain, anxiety, oxytocin, cortisol levels, duration and perception of birth.
  In this regard, the planned targets are;
  * It is to determine the effect of vagus nerve stimulation on labor pain in pregnant women, based on Polyvagal theory.
  * It is to determine the effect of vagus nerve stimulation on the anxiety level of pregnant women, based on the Polyvagal theory.
  * It is to determine the effect of vagus nerve stimulation on the oxytocin level of pregnant women, based on the Polyvagal theory.
  * It is to determine the effect of vagus nerve stimulation on cortisol levels of pregnant women, based on Polyvagal theory.
  * It is to determine the effect of vagus nerve stimulation on the duration of birth of pregnant women, based on the Polyvagal theory.
  * It is to determine the effect of vagus nerve stimulation on the birth perception of pregnant women, based on Polyvagal theory.
Who Masked: Participant
Masking Description: In the study, hormone value analyses, statistics and reporting will be blinded. Before the pre-tests are collected in the collection of data, the responsible researcher will contact the statistician who performed the randomization and reach the randomization list. After learning the group information, the responsible researcher will start the application. The participant will be monitored under the supervision of the responsible researcher until they go to the postpartum care unit. A new participant will be included in the study after the participant is sent to the postpartum care clinic. Therefore, the intervention and control groups will be prevented from seeing each other.
  For hormone analyses, the hormone tubes will be coded as "A" and "B" groups by the responsible researcher. Hormone value analyses will be performed by an expert laboratory technician who is not aware of the groups independent of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): Vagus nerve stimulation based on polyvagal theory and routine application
  Interventions: Other: Vagal Active Tone Application Procedure
- Control Group (No Intervention): Routine maintenance; Routine care and treatment of women will continue during data collection.

INTERVENTIONS:
Other: Vagal Active Tone Application Procedure — First section; A video will be created that includes pictures and visuals describing the vagus nerve, explaining its benefits, and providing information about its effects and usage during the birth process.
  Second section; Deep breathing and focus exercises;
  Feather Breath:
  Candle Breath: The pregnant woman inhaled and exhaled as if she was trying to blow out a candle.
  Relaxation Breath: Deep breath Third section; Body relaxation exercises; Fourth section; Facial muscle relaxation exercises; Fifth section; Neck and larynx muscle relaxation exercises;
  Arms: Intervention Group

SUMMARY:
The vagus nerve innervates both the uterus and the cervix. It is thought that a successful and positive birth experience can be achieved by stimulating the vagus nerve at the desired level. Making instinctive sounds such as singing, humming, and various exercises are methods that stimulate the vagus nerve. In this project, an application protocol based on polyvagal theory and including breathing, relaxation and voice exercises was prepared. Video-supported application material will be developed in line with the prepared protocol. The video-assisted vagus nerve stimulation intervention is called Vagal Active Tone (VAT). VAT is a new method in the literature and for which we have limited information about labor. This project aimed to determine the effect of vagus nerve stimulation based on Polyvagal theory on labor pain, anxiety, oxytocin, cortisol levels, duration and perception of birth. This study was planned as a randomized controlled experimental study. The number of samples was calculated using the G*power 3.1.9.6 program. After the power analysis, it is aimed to reach a total of 50 people, 25 in the intervention group and 25 in the control group. Data will be collected with Personal Information Form, Labor Monitoring Form, Hormone Levels Monitoring Form, Visual Analogue Scale, State Anxiety Scale, Facial Anxiety Scale and Mother's Birth Perception Scale.

It is aimed to produce new and original evidence-based information with the use of VAT intervention based on polyvagal theory. It is thought that this intervention, which can be easily accessed and applied by pregnant women whenever they want, will contribute positively to labor pain, anxiety, oxytocin and cortisol levels, and the duration and perception of birth.

Keywords: Labor, oxytocin, cortisol, vagus nerve stimulation, midwife

ELIGIBILITY:
Inclusion Criteria :

Women who volunteer to participate in the study, are primiparous and in the 28-32nd week of pregnancy, Normal vaginal birth, Single fetus and cephalic presentation, 19 years of age or older, Communicate in Turkish will be included in the study.

Exclusion Criteria:

Women with obstetric complications (placenta previa, preeclampsia, premature rupture of membranes, oligohydramnios, polyhydramnios, presentation disorder, intrauterine growth retardation, İntrauterine dead fetus, macrosomic baby, fetal distress, etc.), Have a psychiatric diagnosis, Have a systemic disease, Have a heart and brain pacemaker, Have epilepsy, Have vision and hearing problems, Attend a childbirth preparation class, Undergo medical procedures for any reason at birth will be excluded from the study.

Ages: 19 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — pregnancy
Enrollment: 50 (Estimated)
Dates: Start 2025-01-25 (Estimated); Primary Completion 2025-03-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) | 30 minutes later (post intervention)
  Visual Analog Scale (VAS): VAS is a one-dimensional scale that objectively evaluates the pain perception of the pregnant woman. It allows some values that cannot be measured numerically to be converted into numerical form. VAS was developed and used by Bond and Pilowsky in 1966. VAS is a 10 cm ruler scale used to quantitatively determine the intensity of pain, with one end representing painlessness (0 = no pain) and the other end representing the most severe pain (10 = severe pain). The patient marks any place between two points that matches the intensity of the pain. The distance between the end of the scale representing painlessness and the point marked by the patient is measured with a ruler and recorded in cm. This numerical value obtained shows the intensity of the pregnant woman's pain.
Facial Anxiety Scale (FAS) | 30 minutes later (post intervention)
  Facial Anxiety Scale (FAS): It is a one-dimensional, individual-based anxiety assessment tool. Its Turkish validity and reliability study was conducted on patients receiving mechanical ventilation in intensive care. Using this numerical rating scale, researchers determined the image corresponding to the patient's facial expression by ranking the face using a number from 0 to 10. A higher score indicates a higher level of anxiety .
State Anxiety Inventory (SAI) | 30 minutes later (post intervention)
  State Anxiety Inventory (SAI): The scale (5) developed by Spielberg and colleagues (1964) to measure the state anxiety levels of normal and abnormal individuals was adapted to Turkish by Öner and Le Compte (1983). The state anxiety inventory was developed to measure a person's anxiety at a certain moment. The 20-item state anxiety inventory is a scale that determines how an individual feels at a certain moment and under a certain condition. SAI is a 4-point Likert-type scale. There are 10 reversed statements on the scale. These statements are items 1, 2, 5, 8, 10, 11, 15, 16, 19 and 20. The state anxiety score is calculated by adding 50 points to the difference between the total weighted scores of direct and reverse statements. The scores obtained in the state anxiety scale theoretically vary between 20 and 80 points. The Cronbach Alpha internal consistency rate of SAI was found to be 0.96.
Maternal Birth Perception Scale (MBS) | 30 minutes later (post intervention)
  Maternal Birth Perception Scale (MBS): It is a tool that assesses how mothers perceive their experiences during normal or unplanned cesarean births. MBS is a 25-item, 5-subscale, and 5-point Likert-type scale developed by Fawcett and Knauth (1997) (7). The sub-dimensions of the scale are experiences during birth (7 items; 3, 5, 6, 8, 15, 17, 18), experiences during the painful period of birth (7 items; 1, 2, 4, 7, 9, 10, 16), postpartum (4 items; 22, 23, 24, 25), spouse participation (4 items; 11,12,20,21), and awareness (3 items; 13,14,19). Since the questions numbered 15-16-17-18-19 of the scale contain negative expressions, the scoring is done in reverse direction in these questions. The translation of ADAÖ into Turkish and the validity and reliability study were carried out by Güngör and Beji (2007). ADAÖ, Cronbach Alpha internal consistency rate was found to be 0.83 (8). Permission for use of the scale was obtained (Appendix-8).
Hormone Values Monitoring Form | 30 minutes later (post intervention)
  Hormone Values Monitoring Form: This is the form in which the oxytocin and cortisol results of the pregnant women participating in the study are monitored.

CONTACTS AND LOCATIONS:
Locations (1):
- Cukurova Unıversıty, Adana, Cukurova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No